CLINICAL TRIAL: NCT01151995
Title: Effectiveness and Costs of Remote Monitoring for Clinical Trials
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Massachusetts General Hospital (Other); University of Michigan (Other)
Responsible Party: Sponsor
Other Study IDs: 09-0735
Record Dates: First submitted 2010-06-24; First posted 2010-06-29 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Remote Monitoring
Keywords: Clinical Trial Monitoring; Effectiveness of remote monitoring; Efficiency of remote monitoring; Costs of remote monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: No biospecimens collected for this protocol
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Remote plus on-site: Subjects will have remote source document verification performed 2-4 weeks prior to study monitors scheduled visit and any variables that were not able to be verified remotely will be verified on-site.
  Interventions: Other: Remote source document verification
- On-site monitoring: Traditional source document verification will be performed when study monitor is on site
  Interventions: Other: On-site source document verification

INTERVENTIONS:
Other: Remote source document verification — Remote access to electronic medical records of the 5 participating sites
  Groups: Remote plus on-site
Other: On-site source document verification — Study monitor will perform on-site source document verification during routine visit to the five participating sites
  Groups: On-site monitoring

SUMMARY:
This pilot project will evaluate Internet-based remote access to electronic clinical systems to support study monitoring tasks. The project engages two NIH-sponsored clinical trial networks (adult: ARDS network; pediatrics: ChiLDREN network) at five trial locations and two coordinating centers located across four states, which engages three collaborating NCRR-funded CTSA institutions. Each study location uses different electronic clinical systems and remote access methods, replicating the diversity of clinical applications and access methods found across large research networks. The results of this pilot project will inform a broader project that will engage all trial sites with electronic clinical systems in both national networks.

This proposal extends Specific Aim 1.2 of the Research Informatics Integrated Core (RIIC) in the parent grant (UL1 RR025780) for the Colorado Clinical and Translational Sciences Institute (CCTSI): "The RIIC will develop and implement tools and services that will….(2) support the efficient execution of the CCTSI translational research projects." (CCTSI grant page 1053). Specific Aim 1.2 proposes to develop new informatics methods that increase the translational research capacity by improving the efficiency of executing clinical studies. Reducing barriers to study monitoring via remote access will enable new innovative approaches to protecting study subjects, ensuring study data quality and documenting regulatory compliance. An example of a completely new model for study monitoring could be continuous study monitoring from any coordinating center to any study location in the Internet-connected world.

We hypothesize that remote monitoring will demonstrate substantial improvements in study monitoring efficiency, effectiveness, and possibly overall costs when compared to present monitoring plans that require a prolonged on-site visit by a study monitor from the coordinating center. We do not claim that remote study monitoring will replace all monitoring tasks . But, for monitoring tasks that require access to electronic clinical data, we seek to demonstrate that remote access can enable more frequent SDV and regulatory documentation compliance, which in turn could facilitate new models of continuous study monitoring. The results of these studies would support improvements in study monitoring that would both significantly reduce the cost of conducting large multi-center clinical while improving the safety of those patients who are enrolled into these trials

DETAILED DESCRIPTION:
II. Research Project Plan Specific Aim 1: To determine the effectiveness of remote access to electronic clinical systems for clinical trial study monitoring. Accuracy and completeness of source document verification (SDV) and compliance with regulatory documentation requirements will be the effectiveness outcome measures.

Specific Aim 2: To determine the efficiency of remote access to electronic clinical systems for clinical trial study monitoring. The time to complete SDV and regulatory review with and without remote access prior to an on-site visit will be the efficiency outcome measures.

Specific Aim 3: To determine the data monitoring site costs of study data verification and regulatory documentation compliance with and without remote access prior to an on-site visit.

Research Methods and Design The specific aims focus on evaluating the effectiveness (Aim 1), efficiency (Aim 2), and cost (Aim 3) of remote study monitoring compared to on-site SDV. The study design for the three Specific Aims is identical. The analysis variables and analytic plan vary by Specific Aim. There are five phases to this project: (1) IT development, (2) local pre-pilot, (3) remote monitoring, (4) on-site monitoring, and (5) study analysis.

Study Phase 1: Initial IT development and testing Five study sites will provide remote access to existing clinical systems using commercial or self-developed access methods. Phase 1 will ensure that these access methods can be configured to provide appropriate security and auditing capabilities. The University of Colorado Hospital (UCH) has identified the need to integrate the McKesson CareManager clinical documentation system into their MedXplore remote access system. The budget provides programming resources to support this integration development during Year 1. Should a technical limitation arise at any location, Phase 1 will be used to alter or extend existing access methods to meet institutional requirements. Contingency plans include using remote desktop sharing, as proposed by Vanderbilt, to export local application screens to remote desktops securely. This contingency ensures that the remote monitor experiences the identical application screens as are seen during on-site visits.

Study Phase 2: Pre-pilot testing of remote monitoring using local study coordinators Study coordinators, local to the five study sites and who have clinical research access privileges already established at their respective hospitals, will perform remote study monitoring review of one or more study subjects to fully test the technical issues of remote access to required applications and the execution features of the data collection instruments. The local coordinators will connect to the hospital systems from a secure computer that is off site from the hospital. The study coordinator will then conduct an on-site chart review. The study coordinator will collect the study measures outlined in Table 2. Procedures for when to stop searching for a data element, how to account for work breaks, and other interruptions, and when to call for additional help from local site managers will be developed. Data collection instruments will be tested and altered as needed. The pre-pilot tests will simulate the activities for Phase 3 & 4 so that all operational issues are resolved. Once completed, study procedures and data collection instruments will be finalized for use in Phases 3 & 4.

Study Phase 3: Remote monitoring by data coordinating centers Randomization of study subjects into two equal arms will be stratified at each individual hospital. Subjects assigned to Arm A will have remote monitoring performed 2-4 weeks prior to the scheduled on-site visit. Subjects assigned to Arm B will have no remote monitoring performed. Both arms will have traditional on-site study monitoring performed. Remote access provisioning performed by IT at the five study locations will allow remote monitors to access electronic records. Depending on institutional responsibilities, HIM or IT resources will provision these remote accounts to access those subjects randomized to Arm A (remote + local monitoring). Remote monitoring will consist of validating all data elements submitted on CRFs submitted to the coordinating center that require source document verification, using the same data verification protocols currently used during on-site visits. Remote monitors will have telephone access to the same HIM and local coordinator resources that are available when on-site. Rules when to stop searching for a data element will be established during Phase 2. Data collection instruments for capturing study variables will be developed and pilot tested during Phase 2. Remote monitors will be trained on the access procedures for each site and the study data collection procedures developed in Phase 2 using simultaneous remote desktop sharing and a study subject who is not scheduled for monitoring.

Study Phase 4: On-site monitoring by data coordinating centers On-site monitoring will occur 2-4 weeks following remote monitoring. Subjects from both Study Arms will have source document verification. Only those elements not verified remotely (Step (A)) will be verified for subjects from Arm A in Step (B). The same monitor will perform both remote and local monitoring for subjects from Arm A. The study variables developed in Phase 2 and used during remote monitoring in Phase 3 will be used during on-site monitoring in Phase 4.

Study Phase 5: Data analysis Specific Aim 1 focuses on accuracy and completeness of remote monitoring versus on-site monitoring. The study variables are the number of variables verified and the number of verified variables that were found to be discrepant. Specific Aim 2 focuses on efficiency, measured in this study as time to complete source document verification and regulatory review. The number of minutes to complete both source document verification and regulatory review will be captured and compared. Specific Aim 3 focuses on costs, measured using a time-in-motion method by the study coordinator or monitor. Using a time log, the time required to complete a CRF to be aggregated for the SDV total. This will include time estimates for finding charts, making copies, and recording data. If a study investigator participates in monitoring activities, then they will record their time estimates separately. Standardized estimates of salaries and benefits for persons in those positions will be used to standardize across local and regional wage and price differentials.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in the NIH-sponsored ARDS and BARC/CLiC clinical trial networks

Exclusion Criteria:

* Not enrolled in the NIH-sponsored ARDS and BARC/CLiC clinical trials

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will be subjects who have already been enrolled in an ARDS or BARC/CLiC clinical trial network study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2010-08; Primary Completion 2010-12 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Effectiveness | 9/2011
  Can remote source document verification replace on-site source document verification?
Efficiency and Cost | 9/2011
  Differences in time and costs

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado at Denver and Health Sciences Center, Aurora, Colorado, United States